CLINICAL TRIAL: NCT05111639
Title: Decision Making for Urinary Diversion in Patients With Bladder Cancer
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Urological Association (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3661.cc; NCI-2021-10463 (Other: CTRP)
Record Dates: First submitted 2021-10-19; First posted 2021-11-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This proposal will aim to improve the understanding about the treatment decision in the type of urinary diversion and identify patient knowledge gaps about uncertainty around patient decision-making.

DETAILED DESCRIPTION:
The Investigator aims to elicit the patient and provider experiences through conducting a 90-minute interview, using an interview guide the research team has developed, using established qualitative research methods for in-depth individual interviews. The team will structure the interviews with broad, open-ended questions to elicit personal thoughts, emotions and experiences regarding decision making for urinary diversion. The team will use the information collected from this interview to make a tool valuable in developing a patient decision aid. For patients who have not undergone surgery yet, the team will ask the patient if it is okay to contact after their surgery to reassess the patients responses to the same questions from the first interview.

In Aim 2, the team will complete part one of the Ottawa decision framework by assessing the patients' and urologists' determinates of decisions for urinary diversion and identify support needs. Using established qualitative research methods for in-depth individual interviews, the team will structure the interviews with broad, open-ended questions to elicit personal thoughts, emotions and experiences regarding decision making for urinary diversion.

Informed by Aim 2 the team will develop a web-based development of a decision aid. The development process will use both the Ottawa decision support and IPDAS to center the design empathetic to the user. The aim will be consistent with principles where the users take priority in the IPDAS guidelines framework and the needs assessment framework. The team will develop a decision support tailored to patients needs who are undergoing urinary diversion and then evaluate the decision making process. The decision aid will use the preferences from the themes of the individual interviews to give patients a preferred method of urinary diversion. The team will perform this in a pre-post fashion.

As mentioned previously, patients will be recruited from the urologists' clinical work. The Indiana and Neobladder patients may have different vantage points in the perioperative period, however at 6-months this should no longer be different. In addition, the team will have patients use the decision aid at 1-month postoperatively to obtain feedback. Getting patient feedback from the group will be critical with such a large number of patients recruited. The research assistant will identify eligible patients prior to their clinic encounter and obtain informed consent. Patients will then complete the decision aid prior to the visit with the surgeon and bring the completed tool into the clinical encounter. After completing the visit, the patient and research assistant will complete the questionnaires assessing acceptability, knowledge, treatment decision and decisional conflict. One month after surgery, our team will also complete the same questionnaires, as well as patient satisfaction and regret at the 6-month follow-up visit. If patients are not available for the visit, our team will attempt to complete telehealth or telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing or who has undergone urinary diversion for bladder cancer
* <90 years old

Exclusion Criteria:

* Any patient undergoing or undergone urinary diversion for other reason than bladder cancer
* aged >90 years old

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants (patients and urologists) will be recruited for qualitative interviews as follows: 1) 10 bladder cancer patients who have undergone urinary diversion within the last year; 2) 10 bladder cancer patients who are undergoing urinary diversion in the next 3 months; and 3) 10 individual interviews will be done with urologists currently performing cystectomy and urinary diversions.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Acceptability of the decision aid tool | 12 months
  Matlock DD, Keech TA, McKenzie MB, Bronsert MR, Nowels CT, Kutner JS. Feasibility and acceptability of a decision aid designed for people facing advanced or terminal illness: a pilot randomized trial.

SECONDARY OUTCOMES:
Knowledge | 12 months
  qualitative analysis of interview data
Decisional Quality | 12 months
  assessed via decisional conflict (Decisional Conflict Scale, O'Connor, 1993 updated 2005), http://www.ohri.ca/decisionaid/
Decisional Regret | 12 months
  Decision Regret Scale, O'connor, 1996, University of Ottawa
Value Concordance | 12 months
  a combination of the above decision quality and regret surveys as well as qualitative analysis of interview data

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kukreja, Principal Investigator — Colorado Research Center
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided